CLINICAL TRIAL: NCT06426056
Title: Nab-Paclitaxel Plus Cisplatin With Concurrent Radiotherapy for Patients With Locally Advanced Cervical Cancer:A Multicentre, Single-arm, Phase II Trial.
Brief Title: Nab-Paclitaxel Plus Cisplatin With Concurrent Radiotherapy for Patients With Locally Advanced Cervical Cancer: A Multicentre, Single-arm, Phase II Trial.
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Jilin Provincial Tumor Hospital (Other); Affiliated Hospital of Hebei University (Other); Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M2024240
Record Dates: First submitted 2024-05-17; First posted 2024-05-23 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-04

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy; Taxes; Paclitaxel; Injections; Cisplatin

STUDY DESIGN:
Intervention Model Description: Radiation Therapy Concurrently With Nab-Paclitaxel Plus Cisplatin
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Image guidance volume modulated arc therapy included 50.4 Gy in 28 fractions to the pelvis and 59.4 Gy simultaneous boost in 28 fractions to involved pelvic and para-aortic lymph nodes, and subsequent high-dose-rate intracavitary brachytherapy at a total dose of 30.0-36.0 Gy in 5-6 fractions, twice a week. Concurrent chemotherapy regimen included weekly cisplatin (40 mg/m^2) and weekly nab-paclitaxel at escalating doses (33 mg/m^2 per week).
  Interventions: Radiation: radiotherapy; Drug: Nab paclitaxel; Drug: Cisplatin

INTERVENTIONS:
Radiation: radiotherapy — Image guidance volume modulated arc therapy included 50.4 Gy in 28 fractions to the pelvis and 59.4 Gy simultaneous boost in 28 fractions to involved pelvic and para-aortic lymph nodes, and subsequent high-dose-rate intracavitary brachytherapy at a total dose of 30.0-36.0 Gy in 5-6 fractions, twice a week.
  Other Names: RT
Drug: Nab paclitaxel — Concurrent chemotherapy regimen included weekly cisplatin (40 mg/m^2) and weekly nab-paclitaxel at escalating doses (33 mg/m^2 per week).
  Other Names: paclitaxel for injection (albumin bound)
Drug: Cisplatin — Concurrent chemotherapy regimen included weekly cisplatin (40 mg/m^2) and weekly nab-paclitaxel at escalating doses (33 mg/m^2 per week).

SUMMARY:
Based on the Phase I trial completed by the sponsor, the Phase II clinical trial aims to investigate the effectiveness and safety of image guidance volume-modulated arc radiation therapy concurrently with Nab-Paclitaxel plus Cisplatin for patients with locally advanced cervical cancer.

ELIGIBILITY:
Inclusion Criteria:

* (1) Stage IB3 to IVA disease based on the 2018 International Federation of Gynecology and Obstetrics (FIGO) system;
* (2) Eastern Cooperative Oncology Group at 2 or less;
* (3) Life expectancy of greater than 3 months;
* (4) Left ventricular ejection fraction at ≥55%;
* (5) Neutrophil count at ≥1500/mm^3, platelet count at ≥100,000/mm^3 or hemoglobin at ≥9.0 g/dL;
* (6) Serum creatinine at <1.5 times the upper limit of the normal reference range;
* (7) Alanine transaminase or aspartate aminotransferase at >2.5 times the upper limit of the normal reference range;
* (8) Non pregnant or lactating women;
* (9) Women of childbearing age willing to adopt reliable contraceptive measures;
* (10) Sign informed consent form.

Exclusion Criteria:

* (1) Individuals who have previously received chemotherapy with albumin bound paclitaxel;
* (2) Individuals who have previously received abdominal or pelvic radiation therapy;
* (3) Individuals who have received neoadjuvant chemotherapy or targeted, immunotherapy, and other anti-tumor treatments prior to concurrent chemoradiotherapy and chemotherapy;
* (4) Individuals with central nervous system diseases or brain metastases；
* (5) Other malignant tumors other than cervical cancer have appeared within the past 5 years;
* (6) Previously experienced sensory or motor neuropathy (Grade ≥ 2) ;
* (7) The researchers evaluate that the uncontrolled serious medical diseases that will affect the ability of the participants to receive the treatment of the clinical trial, such as complicated with serious medical diseases, including serious heart disease, cerebrovascular disease, uncontrolled diabetes, uncontrolled hypertension, uncontrolled infection, active peptic ulcer, etc;
* (8) known to be allergic to paclitaxel;
* (9) Received other experimental drugs or participated in clinical studies for other anti-cancer treatment purposes within 30 days of the first chemotherapy administration;
* (10) Serious infections occurring within 4 weeks prior to the start of research treatment, including but not limited to complications of infection requiring hospitalization, bacteremia, or severe pneumonia;
* (11) Human immunodeficiency virus (HIV) positive individuals;
* (12) Uncontrolled or active viral hepatitis or infection with human immunodeficiency virus;
* (13) Researchers determine that it is not suitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
ORR (objective response rate) | the 1, 3, 6, 9, 12 months after the end of the treatment
  ORR(objective response rate)=CR (complete response)+PR(partial response)/all participants

SECONDARY OUTCOMES:
AE | the 1, 3, 6, 9, 12 months, and 2, 3 years after the end of the treatment
  adverse events
OS | the 1, 2, and 3 years after the end of the treatment
  objective response rate
PFS | the 1, 2, and 3 years after the end of the treatment
  progression-free survival
DOR | the 1, 3, 6, 9, 12 months, and 2, 3 years after the end of the treatment
  duration of response
DCR | the 1, 3, 6, 9, 12 months, and 2, 3 years after the end of the treatment
  disease control rate
CBR | the 1, 3, 6, 9, 12 months, and 2, 3 years after the end of the treatment
  clinical benefit rate

CONTACTS AND LOCATIONS:
Overall Officials: Ping Jiang, Doctor, Principal Investigator — Peking University Third Hospital

IPD SHARING:
Plan to Share IPD: No